CLINICAL TRIAL: NCT06381336
Title: TRAK-SILVER: A Digital Home-Based Physiotherapy Program for Active Aging: a Randomised Controlled Trial.
Brief Title: A Digital Home-Based Physiotherapy Program for Active Aging
Acronym: TRAK-SILVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Collaborators: Basque Health Service (Other Government); University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAKSILVER2022
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Frail Elderly Syndrome; Older Adults
Keywords: telemedicine; active ageing; older people; digital health; pre frail adults; telehealth care

STUDY DESIGN:
Intervention Model Description: A randomized two-group design with pretest-posttest assessment was used to analyse the effectiveness of the TRAK-SILVER application. Seventy-two adults aged 65 and above were stratified by gender and physical functioning capacity (SPBB) and then randomly assigned to either the experimental (EG) or control group (CG). EG received the TRAK-SILVER platform as a treatment methodology. The CG did not have access to the platform and was instructed to continue with the standard care program through exercise sheets.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Use of TRAK-SILVER platform as a treatment methodology.
  Interventions: Device: TRAK-SILVER platform
- Control Group (No Intervention): They did not have access to the platform and were instructed to continue with the standard care program through exercise sheets.

INTERVENTIONS:
Device: TRAK-SILVER platform — The Experimental Group used TRAK-SILVER, a cross-platform web application that empowers healthcare professionals and patients. It facilitates the management of a patient's condition by providing therapeutic exercises, monitoring activity, and administering clinical assessment scales and questionnaires. The platform's advanced artificial vision algorithm, known for its precision, enhances patient engagement with real-time measurements and corrections during exercise.
  Physiotherapists monitored the sessions through the TRAK-SILVER platform's monitoring system and weekly phone calls. The TRAK-SILVER platform had an alert notification system.
  The program's second part involved weekly uploads of health-promoting information pills to the platform.
  Arms: Experimental Group

SUMMARY:
This clinical trial will aim to understand the effects of the TRAK-SILVER digital platform on pre-frail and older adults living at home, assessing its impact on physical activity level, emotional variables, and overall quality of life. Participant satisfaction with the digital treatment will also be evaluated.

This research will provide insight into the utility and acceptance of the digital platform as a personalised and accessible digital physiotherapy program for this population, advancing understanding in the field.

The participants will undergo a 3-month physiotherapy program using the TRAK-SILVER platform or a paper guide based on their assigned group. Additionally, weekly uploads of health-promoting audiovisual content will enhance the intervention's holistic approach to improving older adults' well-being and functional capacity.

DETAILED DESCRIPTION:
The study's recruitment process targets individuals aged 65 and above who live independently in their homes. The social center in Orio, Guipúzcoa, Spain, will serve as a central hub for recruitment. Prospective participants will receive detailed information about the study's requirements, including completing a questionnaire to assess their physical activity levels. They will also be asked to self-report any recent increase in fatigue and weight loss over the preceding month.

After the initial screening, individuals who meet the study's predefined inclusion criteria will be invited to participate. Before enrollment, written informed consent will be obtained from all participants, ensuring ethical compliance and respect for individual autonomy.

The assessment tools used in this study will be comprehensive and systematic, administered both before and after the intervention. The evaluation will cover various metrics, including physical and functional health, mental and emotional well-being, quality of life (QoL), and satisfaction. This approach ensures a thorough evaluation of the intervention's impact on various aspects of the participant's health and well-being.

The study cohort will consist of patients randomly assigned to the experimental group (EG) and the control group (CG). Regardless of group assignment, all patients will undergo baseline health assessments, with the satisfaction questionnaire deferred until post-intervention for both groups.

Participants in the EG will have access to the TRAK-SILVER tool as a fundamental component of the intervention, while participants in the CG will not have such access. Following the intervention phase, which will involve either TRAK-SILVER engagement or adherence to an exercise regimen outlined in a provided sheet, both groups will undergo a new post-intervention assessment, including the satisfaction questionnaire.

The EG will engage in a structured 3-month physiotherapy program comprising 36 60-minute weekly sessions. This program is divided into two distinct phases, each spanning six weeks, with variations in sets and repetitions. Physiotherapists will monitor the sessions using the TRAK-SILVER platform, augmented by weekly phone consultations and email notifications to reinforce engagement.

Each session within the program will include joint mobility exercises, aerobic conditioning, balance training, strength building, and respiratory exercises. Additionally, the platform will feature weekly audiovisual content promoting various aspects of health and well-being to enhance the intervention's efficacy.

In contrast, participants in the CG will receive a printed guide outlining similar recommendations. Adherence to the prescribed regimen will be closely monitored, including session completion rates, post-session pain levels, perceived exertion, and subjective improvement assessments. To enhance adherence, each participant will receive weekly phone calls from supervising physiotherapists.

The study will employ an intention-to-treat analysis approach, incorporating all randomized participants into the final analysis, regardless of their adherence to the intervention protocol. Descriptive statistics, t-tests, and ANCOVA analyses will be utilized to compare changes within and between groups, with statistical significance set at 0.05. Effect sizes will be assessed using Cohen's d.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 65 and living at home (not institutionalized);
* Having a Fried Frailty Index score of 2 points or less.;
* Having a Smartphone, laptop or tablet and having basic knowledge of how to use it or having a person who can help them access and use the platform.

Exclusion Criteria:

* Cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB | up to 3 months
  It is used to classify the participants' physical functioning, with a score below 10 indicating frailty and a high risk of disability or falls.
Gait Speed | up to 3 months
  The Puthoff protocol measured average and maximum gait speed in a six-meter hallway.
Timed Up and Go Test | up to 3 months
  Used to measure the time it took for individuals to stand up from a chair, walk three meters, turn, return to the chair, and sit back down.
6-minute walk test (6MWT) | up to 3 months
  Measure the distance an individual could walk in 6 minutes.
Berg Balance Scale | up to 3 months
  Evaluate balance capacity.
Number of steps count | up to 3 months
  Evaluate walking capacity.
Geriatric Depression Scale-15 (GDS) | up to 3 months
  Assessment mental and emotional well-being. Scores on the GDS range from 0 to 4, indicating the absence of depressive symptoms, while scores from 5 to 8 suggest the presence of mild symptoms.
De Jong Gierveld Loneliness Scale (JGLS) | up to 3 months
  Scores on this scale range from 0 (indicating an absence of loneliness) to 11 (indicating maximum loneliness). To measure the loneliness.
Quality of life (QoL) questionnaire | up to 3 months
  It evaluates health status across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | 3 months
  Client Satisfaction Questionnaire (CSQ), which comprises eight items with four response options, scoring from 8 to 32, with higher scores indicating greater satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Asier Arrizabalaga, Principal Investigator — Zahartzaroa
Locations (1):
- Social Center of Orio (Zahartzaroa), Orio, Basque Country, Spain